CLINICAL TRIAL: NCT06194721
Title: The Effect of Intra-pulpal Anesthesia With Cryotherapy on Intra-operative Pain During Root Canal Treatment on Mandibular Molars With Symptomatic Irreversible Pulpitis
Brief Title: The Effect of Intra-pulpal Anesthesia With Cryotherapy on Intra-operative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Rania Zaarour, Senior Researcher at Thumbay Research Institute Coordinator, Gulf Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-COD-STD-109-JUNE-2023
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Irreversible Pulpitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy (Experimental)
  Interventions: Procedure: Cold intrapulpal anesthesia
- Room temperature (Active Comparator)
  Interventions: Procedure: Room temperature intrapulpal anesthesia

INTERVENTIONS:
Procedure: Cold intrapulpal anesthesia — Intrapulpal cold local anesthesia at 4-5 c temperature
  Arms: Cryotherapy
Procedure: Room temperature intrapulpal anesthesia — Intrapulpal cold local anesthesia at room temperature
  Arms: Room temperature

SUMMARY:
The goal of this clinical trial is to compare the effect of cooling of local anesthesia on intraoperative pain during root canal treatment in mandibular molars diagnosed as symptomatic irreversible pulpitis. The main question it aims to answer is: Is there a difference in intra-operative pain levels using intra-pulpal anesthesia with and without cryotherapy during root canal treatment? Participants will undergo root canal treatment using intrapulpal anesthesia with and without cooling. Researchers will compare cold and room temperature intrapulpal anesthesia to see the intensity of intraoperative pain.

DETAILED DESCRIPTION:
The study will be conducted on 40 mandibular molars in each group n = 20. The patient will be asked to pick an opaque sealed envelope that will contain a number 1 or 2. The resultant number will determine in which group the participants will be placed. Double blinding will be maintained in this study as the assessor and the patients will not be aware of their group.

Group 1: Will receive intrapulpal local anesthesia at 4-5 C after pulp exposure.

Group 2: Will receive intrapulpal local anesthesia at room temperature after pulp exposure.

Procedural steps:

1. A history of present illness will be recorded from the patient and the suspected tooth will be tested for vitality using a cold test and an electric pulp tester, to ensure the correct diagnosis is reached.
2. Once the diagnosis is confirmed to be symptomatic irreversible pulpitis, the patient will receive an inferior alveolar nerve block (2% lidocaine 1:100,000).
3. A rubber dam will be used to achieve isolation, and an access cavity will be prepared using a high-speed handpiece, a round bur (no.4), and an Endo-Z bur.
4. If the patient reports feeling any pain, the procedure will stop, and the patient will be presented with a Visual Analogue Scale and asked to rate the pain on a scale of 1-10. Pain levels of more than 5 will be included in the study.
5. Intra-pulpal anesthesia (2% lidocaine 1:100,000) will be administered, and the needle will be surrounded by a piece of sterile gauze to ensure it is under back pressure.
6. After administering the intra-pulpal injection, the patient will again be presented with the same VAS and asked to rate their current pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mandibular molars diagnosed with symptomatic irreversible pulpitis.
* Mandibular molars with closed apices.
* Patients who are experiencing pain during access cavity drilling above 5 visual analog scale.

Exclusion Criteria:

* • Patients with a known allergy to lidocaine.

  * Root canal-treated mandibular molars.
  * Patients with systemic diseases.
  * Mandibular molars with open apices.
  * Mandibular molars with external/internal resorption.
  * Non-restorable mandibular molars.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-01-06 (Actual)

PRIMARY OUTCOMES:
Level of intraoperative pain | Intraoperative
  Evaluation of intraoperative pain intensity using a visual analog scale. The visual analog scale measures pain intensity. The visual analog scale consists of a 10 cm line, with 2 endpoints representing 0 ( no pain) and 10 (pain as bad it could be)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates